CLINICAL TRIAL: NCT00625079
Title: Randomized Placebo-Controlled Study of Sildenafil For The Treatment of Pulmonary Hypertension Secondary to Idiopathic Pulmonary Fibrosis: A Pilot Study
Brief Title: Pulmonary Hypertension Secondary to Idiopathic Pulmonary Fibrosis And Treatment With Sildenafil
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: inclusion/exclusion criteria limited enrollment
Sponsor: University of California, Los Angeles (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPF/PH
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Arterial Hypertension; Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease; Pulmonary Hypertension
Keywords: pulmonary hypertension; pulmonary arterial hypertension; interstitial lung disease; idiopathic pulmonary fibrosis
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pre-transplant placebo (Placebo Comparator): There are two placebo comparators.... one for the group of patients with resting PAH and another for the group of patients with exercise PAH
  Interventions: Drug: sildenafil
- Pre-transplant sildenafil (Experimental): There are two active comparators, one group with resting PAH and another with exercise PAH, both receiving drug.
  Interventions: Drug: sildenafil
- Pre-transplant no PAH-specific therapy (No Intervention): this group of patients has no evidence for either resting or exercise PAH but will be followed without specific drug intervention

INTERVENTIONS:
Drug: sildenafil — the dose of sildenafil will be 20mg three times per day (orally)
  Other Names: Revatio
  Arms: Pre-transplant placebo; Pre-transplant sildenafil

SUMMARY:
Pulmonary Arterial Hypertension (PAH) in the setting of Idiopathic Pulmonary Fibrosis(IPF)is a risk factor for morbidity and mortality in the peri-lung transplant(LT) setting. Currently there is no significant data to support the use of pulmonary vasodilators for PAH in the setting of interstitial lung disease such as IPF. The majority of IPF patients have PAH either at rest or during exercise. The study hypothesis is that sildenafil may improve morbidity and mortality in the peri-LT setting in both IPF cohorts with either resting or exercise PAH.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the use of sildenafil in patients with pulmonary fibrosis and PH being considered for lung transplantation. We hypothesize that not only will sildenafil improve functionality and QOL in the pre-transplant setting but it may also improve primary graft dysfunction after lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Idiopathic Pulmonary Fibrosis referred for lung transplantation at our medical center
* Minimal 6 minute walk distance of 50 meters; must be able to conduct supine exercise during heart catheterization

Exclusion Criteria:

* Non ambulatory
* Prior adverse reaction/allergy to sildenafil or other PDE-5 Inhibitors
* Any other pulmonary vasodilator within one month of enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
6 minute walk distance (6MWD) change from Baseline | 6 months
  ATS guideline based 6MW distance

SECONDARY OUTCOMES:
Right heart catheterization hemodynamics | initial right heart catheterization compared to catheterization done on day of lung transplantation; we will specifically compare mean pulmonary artery pressure, pulmonary vascular resistance, and pulmonary artery wedge pressure
  pulmonary hemodynamics via invasive right heart catheterization
Chemokine analysis on peripheral blood | the chemokines will be quantified and compared between study entry and the time point just prior to lung transplantation
  evaluation of a group of chemokines before and after the intervention in each arm
Quality of life assessment | study entry compared to 6 months or at the time of lung transplantation (whichever comes first); there is a 0-100 scoring scale and the lower the score, the more disability
  SF-36 (short-form 36)
Quality of life assessment in the context of dyspnea | the SGRQ will be be compared at two time points, study entry and at 6 months or the time of transplantation (whichever comes first); scores range from 0 to 100 and higher scores indicate more limitation
  Saint George Respiratory Questionnaire (SGRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Rajan Saggar, MD, Study Director — David Geffen School of Medicine, UCLA
Locations (1):
- David Geffen School of Medicine UCLA, Los Angeles, California, United States